CLINICAL TRIAL: NCT03370419
Title: The Pick Two to Stick To Habit Development Intervention
Acronym: P2S2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Heather Fritz, Assistant Professor of Occupational Therapy and Gerontology, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1601014563
Record Dates: First submitted 2017-12-04; First posted 2017-12-12 (Actual); Results first posted 2019-12-02 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2019-11

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Habits; African American; Emergency Medicine
MeSH Terms: conditions — Metabolic Syndrome; Habits | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Two group randomized controll trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Pick Two to Stick To (Experimental): Participants are asked to participate in five health-coaching sessions and to return in Week 20 for follow-up data collection. The initial face-to-face coaching session lasts approximately 90 minutes with subsequent telephone sessions lasting approximately 20 minutes. Coaching sessions will include education about MetS, weight loss, dietary and physical activity recommendations, and the principles of habit development, guidance in forming implementation intentions for each self-selected habit, and identifying routines and contextual cues that could be modified to support habit development Coaching sessions are augmented with a participant workbook. Participants' also receive individually tailored study text messages to maintain their motivation.
  Interventions: Behavioral: Treatment
- Usual Care (Other): Participants receive usual care only.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Treatment — Lifestyle intervention fostering the development of behavioral automaticity (habit strength) or dietary and physical activity behaviors.
  Arms: The Pick Two to Stick To
Behavioral: Usual care — Usual care
  Arms: Usual Care

SUMMARY:
Metabolic syndrome (MetS) is a leading risk factor for chronic disease among African American/Black populations. Fostering habit development offers a promising new approach to improving the effectiveness of lifestyle programs for people with MetS, yet this approach remains understudied. The long-term goal of this line of research is to test and disseminate an affordable and effective intervention for reducing MetS. The objective of the proposed project is to evaluate the feasibility of a novel, occupational therapist-delivered habit-development intervention targeting dietary and physical activity habits in up to 100 African American/Blacks with MetS ages 40+ recruited from an emergency department in Detroit, MI. The specific aims are to (a) evaluate intervention feasibility and acceptability and (b) estimate intervention effect sizes for primary outcome measures of habit development and weight loss and secondary outcomes of blood pressure, BMI, and waist circumference. Through the 8-week intervention, indicators of intervention feasibility (e.g., time, effort, costs, participant recruitment and retention, satisfaction) will be tracked. Measures of habit development will be taken biweekly over the 8-week active intervention period and anthropometry measures will be collected at baseline and week 20.

DETAILED DESCRIPTION:
Together, diabetes and cardiovascular disease cost the U.S. economy a staggering $557.6 billion annually and are the leading chronic diseases of African Americans. Maintaining a healthy body weight by being physically active and eating a healthy diet are the best means of reducing cardio-metabolic risk factors. Despite decades of behavioral research, however, lifestyle interventions targeting activity and diet have made little progress in effecting widespread and enduring health behavior changes in the populations most at risk for developing these conditions. Addressing the role of habits, defined as behavior patterns operating below conscious awareness that are acquired through context-dependent repetition, would significantly improve the effectiveness of lifestyle interventions. Most simply, habits develop when repetition of a behavior (e.g., walking for 10 minutes) occurs in connection with a stable situational cue that supports the behavior (e.g., while on a lunch break). Once established, habits are cued by the characteristics of a specified recurring situation rather than by intentions. Recent research suggests that habit development may prevent relapse and aid maintenance of behavior changes beyond the duration of the intervention because the performance of habitual behaviors is less vulnerable to changes in motivation, mood, or extraneous circumstances. Emerging evidence also suggests that habit-development strategies are (a) effective across a range of behaviors (e.g., dental flossing, physical activity, and dietary behaviors); (b) effective in low doses; and (c) deliverable via multiple formats (e.g., paper or electronic). Such strategies could therefore be feasibly implemented in a range of settings to target the development of healthful physical activity and dietary habits. Nonetheless, these concepts and methods have yet to be fully tested to determine their feasibility as a treatment modality for promoting healthful lifestyle behavior changes.

The long-term goal of the larger research project of which this is a part is to disseminate an affordable and effective intervention adaptable to a variety of healthcare settings for fostering healthful physical activity and dietary habits, thereby reducing the burden of related chronic diseases on affected individuals and society. The short-term objective of the proposed research is to test the feasibility of a habit-focused intervention in a sample of 80 African American adults ages 40 and older with metabolic syndrome (MetS). The overarching hypothesis is that a habit-focused approach will be feasible to implement and acceptable to intervention recipients. Rooted in habit theory and informed by the information-motivation-behavioral (IBM) model, the brief 8-week intervention consists of one face-to-face consultation, four bi-weekly individual tele-coaching sessions, and the use of ambulatory momentary assessments (via a smartphone application) to support the development of healthy dietary intake and physical activity habits and improve key health outcomes. The two specific aims of the study are:

1. To evaluate intervention feasibility and acceptability. Determine if the intervention used in the proposed project is feasible. By tracking time, effort, costs, adherence to recommendations, participant recruitment and retention rates, and intervention satisfaction, it is expected that we will obtain data that both support the feasibility of the intervention and help improve it for a subsequent study.
2. To estimate intervention effect sizes for the primary outcome measures of habit development and for the secondary outcome measures of blood pressure, BMI, and waist circumference. Habit development and anthropometry will be measured using the four-item Self-Reported Behavioral Automaticity Index (Gardner et al., 2012) biweekly during the active intervention, weeks 2, 4, 6, and 8.

ELIGIBILITY:
Inclusion Criteria

* Two of the following three MetS risk factors (waistline > 40 inches for men and > 35 inches for women; blood pressure > 130/85; HbA1c of 5.7%-6.4%)
* Adults who present to the ED with non-life threatening conditions
* English-speaking subjects who will be discharged to home from the ED

Exclusion Criteria:

* Pregnant patients
* Previous diagnosis of resistant HTN
* Steroid-dependent asthma or emphysema
* Cirrhosis or hepatic failure
* Cardiac event within the last 30 days
* Chronic kidney disease on renal replacement therapy
* Cancer (terminal or undergoing active chemotherapeutic or radiation therapy)
* Taking medications for weight reduction or already being involved in a weight reduction program.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Fritz, PhD, Principal Investigator — Wayne State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fritz H, Tarraf W, Brody A, Levy P. Feasibility of a behavioral automaticity intervention among African Americans at risk for metabolic syndrome. BMC Public Health. 2019 Apr 16;19(1):413. doi: 10.1186/s12889-019-6675-7. PMID 30991972

RESULTS

PARTICIPANT FLOW:
Groups:
- The Pick Two to Stick To: Participants are asked to participate in five health-coaching sessions and to return in Week 20 for follow-up data collection. The initial face-to-face coaching session lasts approximately 90 minutes with subsequent telephone sessions lasting approximately 20 minutes. Coaching sessions will include education about MetS, weight loss, dietary and physical activity recommendations, and the principles of habit development, guidance in forming implementation intentions for each self-selected habit, and identifying routines and contextual cues that could be modified to support habit development Coaching sessions are augmented with a participant workbook. Participants' also receive individually tailored study text messages to maintain their motivation.
  The Pick Two to Stick To Habit Development Intervention: Lifestyle intervention fostering the development of behavioral automaticity (habit strength) or dietary and physical activity behaviors.
  Control: usual care
Period: Overall Study
Arm/Group | The Pick Two to Stick To
Started | 40
Completed | 24
Not Completed | 16
Not completed — Lost to Follow-up | 16

BASELINE CHARACTERISTICS:
Arm/Group | The Pick Two to Stick To
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 49 [40 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 40
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Behavioral Automaticity Index
Description: Habit strength, operationalized as changes in behavioral automaticity, were measured using a 1-7-point Likert scale. Participants respond to 4 stem statements. The scale thus ranges from 4-28. Higher score indicated a stronger habit.
Time Frame: 2 weeks
Population: 12 of the 24 participants who entered the trial dropped and as such there was only complete data on 12 participants.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | The Pick Two to Stick To
Number analyzed (Participants) | 12
score on a scale | 10.4 (0.4)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | The Pick Two to Stick To
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-01-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT03370419/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-07-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT03370419/Prot_SAP_001.pdf